CLINICAL TRIAL: NCT03825185
Title: Transsternal Versus Transcervical Thymectomy for the Management of Myasthenia Gravis: A Randomized Controlled Trial With a Mean Follow-up of 10 Years
Brief Title: Transsternal Versus Transcervical Thymectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBH 531 (1995)
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Myasthenia Gravis, Thymectomy
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: A total of 100 patients with diagnosis of MG referred to our center for surgical treatment between 1993 and 2003 were invited to participate in the study. Software (Power and Precision, Biostat, NJ) was used for sample size calculation. Software (G* Power 3.1) was used for sample size calculation. Sample size was calculated based on a 4.0% difference in the remission rate between TC (40%) and TS (44%). The calculated sample size was 26 patients in each group. Considering a 10 to 20% loss of follow up in the long term, a total of 50 patients per group were included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcervical Thymectomy (Experimental): 50 patients were randomized to transcervical thymectomy for treatment of myasthenia gravis.
  Interventions: Procedure: Transcervical Thymectomy
- TranssternalThymectomy (Experimental): 50 patients were randomized to transternal thymectomy for treatment of myasthenia gravis.
  Interventions: Procedure: Transsternal Thymectomy

INTERVENTIONS:
Procedure: Transcervical Thymectomy — Transcervical Thymectomy. All transcervical thymectomies were performed with an 8 cm transversal cervicotomy was performed approximately 2 cm above the sternal notch. Musculocutaneous flaps were developed up to the thyroid cartilage and the suprasternal notch. Strap muscles were split in the middle and retracted laterally. The upper horns of the thymus were exposed and were freed up to the level of the innominate vein. All tributary veins were suture ligated. A sternal retractor was then placed to retract the sternum upward until the patient was nearly lifted off the table. The rest of the Thymus was dissected, from the pericardium and the pleura. Care was specially taken to remove as much fatty tissue adjacent to the thymus as possible preserving the phrenic nerves.
  Arms: Transcervical Thymectomy
Procedure: Transsternal Thymectomy — Transsternal Thymectomy. A standard formal median sternotomy was carried out. The sternum was retracted laterally using an automatic retractor. All thymic tissue with the adjacent adipose tissue was removed starting with the inferior horns of the thymus. Thymic vessels were ligated and dissection was continued until the upper horns could be separated from the thyroid. A mediastinal tube was placed before closing the sternum and was kept in close suction for 2 to 3 days.
  Arms: TranssternalThymectomy

SUMMARY:
Objective: To comparatively analyze long-term results and complications of transcervical (TCT) and transsternal thymectomy (TST) in a randomized controlled trial with a mean follow-up of ten years.

Results: Outcomes 10 years after surgery by MGFA post-intervention status showed that complete stable remission was achieved in 8 (21.6%) patients of the TCT group, and in 20 patients (55.5%) of the TST group.

Conclusions: Transcervical and transsternal thymectomy are safe and result in significant improvement of patients with Myasthenia Gravis. TST has superior results in terms of complete stable remission at 10 years.

DETAILED DESCRIPTION:
Background: Thymectomy is an effective treatment for Myasthenia Gravis in the adult population. Surgical removal of the thymus can be performed through several approaches. Comparison of the most commonly used surgical techniques through randomized control trials with long-term follow-up is scarce.

Objective: To comparatively analyze long-term results and complications of transcervical (TCT) and transsternal thymectomy (TST) in a randomized controlled trial with a mean follow-up of ten years.

Results: A total of 100 patients were randomized to transsternal thymectomy (50), and transcervical procedure (50). There were not significant differences in the demographic characteristics, MGFA clinical classification, and MGFA therapy status between groups before surgery. Twenty patients were lost of follow up during the first year and were excluded. Our final group included 40 patients in each group. Three patients in TCT group (7.5%) and 6 patients in the TST group (15%) developed surgical complications. At 1 year of follow-up, 7 patients (17.5%) of the TCT group were asymptomatic in comparison with 15 patients (37.5%) of group TST, after 10 years of follow-up, 26 cases (72.9%) in group TCT were asymptomatic in comparison with 29 cases (80.5%) of group TST. Outcomes 10 years after surgery by MGFA post-intervention status showed that complete stable remission was achieved in 8 (21.6%) patients of the TCT group, and in 20 patients (55.5%) of the TST group.

Conclusions: Transcervical and transsternal thymectomy are safe and result in significant improvement of patients with Myasthenia Gravis. TST has superior results in terms of complete stable remission at 10 years.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were a clinical diagnosis of MG confirmed by biochemical or physiologic studies and a CT excluding thymoma. -

Exclusion Criteria:

Exclusion criteria were contraindications for major surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 1993-01-01 (Actual); Primary Completion 2004-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pharmacological remission of MG. | 10 years
  Remission of MG classified according to MGFA Post intervention status for postoperative remission of Myasthenia Gravis
Clinical remission of MG. | 10 years
  Remission of MG classified according to MGFA Post intervention status for postoperative remission of Myasthenia Gravis
Pharmacological and clinical remission of MG. | 10 years
  Remission of MG classified according to MGFA Post intervention status for postoperative remission of Myasthenia Gravis

IPD SHARING:
Plan to Share IPD: No